CLINICAL TRIAL: NCT07130240
Title: Ivonescimab Combined With Paclitaxel and Cisplatin as Neoadjuvant Therapy Followed by Type A Hysterectomy in Stage IB2 and IIA1 Cervical Cancer: A Phase II Trial
Brief Title: Ivonescimab Combined With Paclitaxel and Cisplatin as Neoadjuvant Therapy Followed by Type A Hysterectomy in Stage IB2 and IIA1 Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Keqin Hua, Director of gynecological oncology, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YIWX-CER-001
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant Ivonescimab combined with paclitaxel and cisplatin (Experimental): Drug: Neoadjuvant Chemotherapy paclitaxel, 135-175mg/m2, q3w, 2-3 cycles
  Drug: Neoadjuvant Chemotherapy cisplatin, 75-80mg/m2, q3w, 2-3 cycles
  Drug: Immunotherapy Ivonescimab, 20mg/kg, q3w, 2-3cycles
  Procedure: Type A hysterectomy After 2-3 cycles of neoadjuvant therapy, patients who achieve CR/PR (evaluated by MRI) and meet SHAPE criteria will receive Type A hysterectomy plus sentinel lymph node dissection / pelvic lymphadenectomy
  Interventions: Drug: Neoadjuvant Chemotherapy Combined with Immunotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy Combined with Immunotherapy — Drug: Neoadjuvant Chemotherapy paclitaxel, 135-175mg/m2, q3w, 2-3 cycles
  Drug: Neoadjuvant Chemotherapy cisplatin, 75-80mg/m2, q3w, 2-3 cycles
  Drug: Immunotherapy Ivonescimab, 20mg/kg, q3w, 2-3cycles
  Procedure: Type A hysterectomy After 3 cycles of neoadjuvant therapy, patients who achieved CR/PR will undergo Type A hysterectomy + sentinel lymph node dissection / pelvic lymphadenectomy

SUMMARY:
Cervical cancer ranks fourth globally in both incidence and mortality rates, making early diagnosis and treatment of great significance. For early-stage cervical cancer, surgery remains the primary treatment approach. According to the latest NCCN guidelines, patients with Stage IA2 or IB1 cervical cancer confirmed by cone biopsy who meet Concerv or SHAPE criteria no longer require type C/B hysterectomy. Instead, they may undergo type A hysterectomy with reduced surgical margins. However, patients with Stage IB2 or IIA1 tumors measuring 2-4 cm still require radical hysterectomy (type C). Radical hysterectomy carries high risks of postoperative complications and significantly impairs quality of life, including major vascular injury, urinary tract damage and dysfunction, lymphatic complications, and sexual dysfunction. Therefore, there is an imperative need to explore alternative or refined treatment approaches for Stage IB2/IIA1 cervical cancer that ensure survival outcomes while reducing surgical morbidity and improving quality of life.

Neoadjuvant therapy followed by scale-reduced surgery may represent a feasible strategy. Both immune escape and angiogenesis are core drivers of tumorigenesis and progression. Combined immunotherapy and anti-angiogenic therapy have demonstrated favorable antitumor efficacy and manageable safety profiles across multiple tumor types. Ivonescimab is a novel humanized tetrameric IgG-scFv bispecific antibody targeting PD-1 and VEGF. Mechanistically, PD-1 blockade reverses T-cell suppression while VEGF inhibition curbs neovascularization, yielding synergistic therapeutic enhancement. This agent has shown promising efficacy and safety in advanced non-small cell lung cancer, hepatocellular carcinoma, and recurrent glioblastoma, though clinical data in cervical cancer remain absent. Therefore, this prospective exploratory study aims to evaluate the efficacy and safety of neoadjuvant Ivonescimab combined with paclitaxel and cisplatin followed by type A hysterectomy for stage IB2/IIA1 cervical cancer. The findings may provide novel insights for optimizing treatment paradigms-ensuring survival outcomes while preserving quality of life.

DETAILED DESCRIPTION:
Cervical cancer, one of the three major malignancies of the female reproductive system, poses a significant threat to women's health. According to global cancer statistics, it ranks as the fourth most common cancer in women. The latest NCCN guidelines indicate that early-stage cervical cancer patients meeting SHAPE criteria (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma; FIGO 2009 stage IA2 or IB1; tumor size ≤2 cm; stromal invasion depth <10 mm on LEEP/cone biopsy or <50% on MRI; any histological grade; no lymph node metastasis) may undergo type A hysterectomy. However, patients with Stage IB2 or IIA1 disease (2 cm < lesion size ≤4 cm) still require radical hysterectomy (type C). Compared to type A hysterectomy, radical hysterectomy carries higher postoperative complication rates and significantly impairs quality of life, including risks of major vascular injury, urinary tract damage and dysfunction, lymphatic complications, and sexual dysfunction. Therefore, there is an urgent need to develop alternative or refined treatment approaches for Stage IB2/IIA1 cervical cancer that ensure survival outcomes while improving quality of life and reducing complications associated with extensive radical surgery.

In recent years, immunotherapy has emerged as a major research focus in oncology. Anti-PD-1/PD-L1 monoclonal antibodies, as immunotherapeutic agents, have demonstrated favorable antitumor efficacy and manageable toxicity in clinical trials. PD-1, a surface immune checkpoint protein, inhibits T-cell activation upon binding to its ligand PD-L1, enabling tumor immune evasion. The NACI study investigated neoadjuvant chemotherapy combined with camrelizumab for locally advanced cervical cancer. Promising results showed an ORR of 98% (83/85, 95% CI: 98%-100%) in the overall population (n=85), with 16 patients (19%) achieving complete response (CR) and 67 (79%) partial response (PR). The pathological complete response (pCR) rate was 38% (32/85, 95% CI: 27%-49%), demonstrating significant clinical benefit with controllable safety, thus ushering in a new era for cervical cancer neoadjuvant therapy. Additionally, a phase II clinical trial reported at the 2024 ASCO Annual Meeting evaluated sintilimab combined with paclitaxel and cisplatin as neoadjuvant therapy for locally advanced cervical cancer, showing a pCR rate of 32.6% (14/43) and an optimal response rate (residual tumor depth <3 mm) of 51.2% (22/43). Regarding toxicity, 15 patients experienced grade 3-4 neutropenia without other severe adverse events, indicating favorable antitumor activity and manageable toxicity for this combination approach. These findings raise the question: Could this immunotherapy-chemotherapy strategy be applied to earlier-stage disease-specifically neoadjuvant treatment for Stage IB2/IIA1 cervical cancer-potentially enabling surgical de-escalation?

Bevacizumab plus chemotherapy constitutes the standard first-line treatment for metastatic or recurrent cervical cancer. Angiogenesis plays a pivotal role in tumor progression by supplying nutrients and oxygen, facilitating tumor growth and dissemination, and remodeling the tumor microenvironment. The phase 3 BEATcc trial published in The Lancet demonstrated that adding atezolizumab (a PD-L1 inhibitor) to standard care (bevacizumab + chemotherapy) significantly improved progression-free survival (PFS) and overall survival (OS) in metastatic, persistent, or recurrent cervical cancer, providing clinically meaningful benefits and suggesting superior efficacy with combined anti-angiogenic and immunotherapy. Another 2024 ASCO report from a randomized phase III trial (NCT04678791) showed that nimotuzumab (an anti-EGFR mAb) combined with concurrent chemoradiotherapy significantly improved ORR in locally advanced cervical cancer, with favorable trends in PFS/OS and an acceptable safety profile. The nimotuzumab group achieved partial response (PR) in 62 patients (43.99%) and complete response (CR) in 57 (40.14%), highlighting the clinical value of anti-angiogenic therapy combined with chemotherapy for locally advanced disease. Given that both angiogenesis and immune escape contribute to treatment resistance, could dual-pathway targeting yield synergistic (1+1>2) effects? However, no studies have yet explored combined anti-angiogenic and immunotherapy as neoadjuvant treatment for Stage IB2/IIA1 cervical cancer.

Ivonescimab, a humanized anti-PD-1/VEGF bispecific antibody with an IgG1-scFv tetrameric structure, represents a novel therapeutic format. As the world's first PD-1/VEGF bispecific antibody to enter phase III trials, it has now gained approval. At the 2024 ASCO meeting, ivonescimab combined with platinum-doublet chemotherapy demonstrated robust antitumor activity and safety not only in first-line treatment of advanced NSCLC without driver mutations but also in EGFR-mutant patients after EGFR-TKI failure and in platinum/PD-(L)1 inhibitor-pretreated advanced NSCLC. This suggests significant efficacy of bispecific antibodies in advanced malignancies. Therefore, given the unmet need for optimized therapies in Stage IB2/IIA1 cervical cancer, this study will explore the efficacy and safety of neoadjuvant ivonescimab combined with paclitaxel and cisplatin. The findings may enable subsequent surgical de-escalation to type A hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

(1)Patients with FIGO 2018 stages IB2, IIA1 (2< lesion ≤4 cm, confirmed by MRI); (2) Histologically confirmed cervical squamous cell carcinoma, cervical adenocarcinoma, or cervical adenosquamous carcinoma; (3)18-75 years old. (4) ECOG performance status score: 0-1. (5) No prior therapy received by the participant. (6)Expected survival period ≥6 months. (7) Women of childbearing potential must agree to use contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the study and for 6 months after the study ends. A negative serum or urine pregnancy test within 7 days before study enrollment is required, and the patient must not be breastfeeding.

(8) Adequate organ function as defined by the protocol, with test samples collected within 7 days before the start of study treatment.

(9) Participants voluntarily join the study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Histological subtypes or disease stages other than those permitted in inclusion criteria (1) and (2).
2. Severe hypersensitivity (≥ Grade 3) to cisplatin, paclitaxel, Ivonescimab , and/or any of their excipients.
3. Participation in another clinical trial within 4 weeks prior to enrollment.
4. Administration of inactivated vaccines within 30 days before the first study treatment or planned vaccination during the study period.
5. Treatment with systemic immunostimulants, colony-stimulating factors, interferons, interleukins, or combination vaccines within 6 weeks or 5 half-lives (whichever is shorter) before the first dose.
6. Diagnosis of immunodeficiency or chronic systemic steroid therapy (exceeding 10 mg prednisone equivalent per day) or any other form of immunosuppressive therapy within 7 days before the first dose.
7. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressive drugs) within the past 2 years.
8. History of (non-infectious) pneumonitis requiring steroid treatment or current (non-infectious) pneumonitis.
9. Active infection requiring systemic treatment.
10. Known history of HIV infection.
11. Known history of hepatitis B (defined as HBsAg reactivity) or active hepatitis C virus infection (defined as detectable HCV RNA [qualitative]).
12. Known history of active tuberculosis (TB; Mycobacterium tuberculosis).
13. Prior allogeneic tissue/solid organ transplantation.
14. Central nervous system metastases, such as brain metastases.
15. Uncontrolled pleural or peritoneal effusion.
16. Impaired mobility due to pathological fractures caused by bone metastases.
17. Insufficient bone marrow function (without transfusion within 14 days): a) Absolute neutrophil count (ANC) <1.5×10⁹/L;b) Platelets <100×10⁹/L; c) Hemoglobin <9 g/dL.
18. Liver abnormalities: a) ALT, AST, or ALP >2.5× upper limit of normal (ULN) without liver metastasis or >5×ULN with liver metastasis; b) Total bilirubin >1.5×ULN (>3×ULN in patients with Gilbert's syndrome); c) Decompensated cirrhosis (Child-Pugh class B or C); d) HBsAg-positive with HBV DNA ≥2000 IU/mL (patients with HBsAg-positive and HBV DNA <2000 IU/mL must receive at least 2 weeks of anti-HBV therapy before the first dose); e) HCV antibody-positive with detectable HCV RNA.
19. Kidney abnormalities: a) Serum creatinine >1.5×ULN or estimated creatinine clearance <60 mL/min using the Cockcroft-Gault formula; b) Urinalysis showing protein ≥++ and confirmed 24-hour urine protein >1.0 g; c) Renal failure requiring hemodialysis or peritoneal dialysis; d) History of nephrotic syndrome.
20. Bleeding risk: a) Coagulation abnormalities: Activated partial hromboplastin time (APTT) or thrombin time (TT) >1.5×ULN, or international normalized ratio (INR) >1.5 (>2.5 for patients requiring anticoagulation therapy); b) History of bleeding (e.g., hemoptysis), coagulation disorders, or current use of warfarin, aspirin, low-molecular-weight heparin, or other antiplatelet agents (except for aspirin ≤100 mg/d for prophylaxis); c) Any signs or history of bleeding diathesis, regardless of severity; d) Active gastrointestinal bleeding, evidenced by hematemesis, hematochezia, or melena within the past 3 months, without resolution confirmed by endoscopy or colonoscopy; e) Any CTCAE ≥ Grade 3 bleeding or hemorrhagic event within 4 weeks before the first dose.
21. Cardiovascular and cerebrovascular abnormalities: a) Any of the following within 12 months before the first dose: ≥ Grade 2 myocardial ischemia, yocardial infarction, arrhythmias, ≥ Grade 3 cardiac insufficiency, uncontrolled angina, coronary/peripheral artery bypass graft surgery, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack; b) Deep vein thrombosis or pulmonary embolism within 6 months before the first dose; c) Left ventricular ejection fraction (LVEF) <50% assessed by Doppler ultrasound; d) Average QTc interval corrected by Fridericia's formula (QTcF) (based on at least 3 consecutive ECG readings): ≥470 ms for females; e) Uncontrolled hypertension (at least 2 measurements showing systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
22. Other factors judged by the investigator as potentially affecting study results or leading to premature termination, such as alcoholism, drug abuse, other severe diseases (including mental illness) requiring concurrent treatment, significant laboratory abnormalities, or family/social factors that may compromise patient safety.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6-9 weeks
  ORR measures the proportion of patients whose cervical cancer shows a complete response (CR) or partial response (PR) to neoadjuvant therapy in this study. Complete Response (CR) means total disappearance of all detectable tumors and partial Response (PR) means significant reduction in tumor size larger than 30% according to RECIST guidelines.
Pathological Complete Response (pCR) | 3 months
  Pathological Complete Response (pCR) refers to the absence of detectable cancer cells in the tissue removed during surgery after neoadjuvant therapy which is examined under a microscope by a pathologist.

SECONDARY OUTCOMES:
OS (Overall Survival) | 2 years
DFS (Disease Free Survival) | 2 years
Adverse Events | 2 years
Changes in tumor-related biomarkers | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Obstetrics & Gynecology Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No